CLINICAL TRIAL: NCT07165379
Title: Analysis of Neuromodulation as a Complementary Treatment to Evidence-based Clinical Intervention in Subjects With Musculoskeletal Pathology of the Lower Limb: a Double-blind Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Manuel González-Sánchez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151/2025
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Neuromodulation; Lower Limb; Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neuromodulation 2 times per week (Experimental)
  Interventions: Other: Neuromodulation; Other: Physical Exercise; Other: Stretching
- Neuromodulation 3 times per week (Experimental)
  Interventions: Other: Neuromodulation; Other: Physical Exercise; Other: Stretching
- Non-neuromodulation 2 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching
- Non-neuromodulation 3 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching

INTERVENTIONS:
Other: Neuromodulation — The application of neuromodulation therapy will be carried out with the support of ultrasound visualization on the anatomical area of the target nerve, seeking a motor and/or sensory response with its stimulation.
  Arms: Neuromodulation 2 times per week; Neuromodulation 3 times per week
Other: Physical Exercise — The therapeutic physical exercise will consist of 3 periods of isometric contraction of 30 seconds, with a rest period of 1 minute, varying the number of repetitions from 3 to 5 depending on the patient's symptoms.
Other: Stretching — To stretch the muscles involved, perform three periods of maximum tolerable stretching without pain, lasting 20 seconds and resting for 30 seconds.

SUMMARY:
This project aims to analyze the use of neuromodulation within a treatment protocol for musculoskeletal conditions of the lower limb, as well as to determine the difference between two and three sessions per week. Study participants will be divided into four intervention groups: the first will receive two sessions per week for a period of six months, while the second will receive three sessions per week for the same period. The treatment protocol will consist of therapeutic physical exercise focused on the muscles and joints of the lower limb, stretching of the involved muscles, and neuromodulation of the nerve root of the lumbosacral plexus, which innervates the affected structures. The third and fourth intervention groups will receive the same treatment as mentioned above, but without neuromodulation. The third group will receive three sessions per week, while the second group will receive two sessions per week. Two different types of measurement variables will be used: objective variables will be used to measure range of motion and muscle strength. Subjective variables will also be used through validated questionnaires, covering physical activity, health-related quality of life, lower limb function, and a visual analog scale for pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study will be men and women of working age, diagnosed with musculoskeletal disorders of the lower limb, and who have not yet received physical therapy.

Exclusion Criteria:

* Have undergone surgery.
* Those who refuse to participate in this study.
* Patients who present muscular atrophy in the lower limb due to a pathology of the latter.
* Medical conditions that are contraindications for neuromodulation therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
EUROQOL-5D (EQ-5D) | Baseline and up to one year
  It consists of a generic instrument for measuring health-related quality of life (HRQoL), which consists of two parts: a descriptive system for assessing health status (ranging from 1, meaning "I have no problems" to 3, "many problems") and a visual analogue scale (ranging from 0, which is the worst imaginable health status, to 100, which is the best imaginable health status).
SHORT FORM 12 HEALTH SURVEY (SF-12) | Baseline and up to one year
  The SF-12 questionnaire is composed of a subset of 12 items derived from the SF-36, with the physical and mental components being scored as the only items. Depending on the item, response options range from 3 to 6, with each question receiving a value that is subsequently transformed into a scale of 0 to 100. All scores have a mean of 50, with values above or below 50 indicating better or worse health status, respectively, compared to the reference population.
LOWER EXTREMITY FUNCTIONAL SCALE (LEFS) | Baseline and up to one year
  This questionnaire assesses perceived functionality in patients with a musculoskeletal problem in the lower limb. It consists of 20 questions, each of which is scored by the patient, ranging from 0 (extreme difficulty or inability to perform the activity) to 4 (no difficulty). The maximum score is 80 (no functional limitations), and the minimum score of 0 indicates extreme limitation. The Spanish adaptation has demonstrated similar values to the English version in the areas of internal consistency, reliability, structure, and error.
LOWER LIMB FUNCTIONAL INDEX (LLFI) | Baseline and up to one year
  This is a 25-item questionnaire that measures lower extremity function. Patients are asked to answer YES if they can perform the action (1 point) and NO if they cannot (0 points). There is also a HALF option (partially able to perform it), which is worth 0.5 points. The score is then obtained by summing the responses and is finally converted into a 100-point percentage scale.
International Physical Activity Questionnaire (IPAQ) | Baseline and up to one year
  An instrument designed to measure physical activity levels in an adult population and serve as a reference for making recommendations regarding physical activity. It comes in two versions: the long version with 31 items (IPAQ-LF) and the short version with 9 items (IPAQ-SF). The short version, which will be used in this study as recommended by the authors, measures activity at four intensity levels, ranging from 1 (vigorous activity) to 4 (sedentary).
Visual Analogue Scale (VAS) | Baseline and up to one year
  It consists of an 11-point numerical scale, ranging from 0 (no pain) to 10 (maximum pain intensity), which serves as a quantification for measuring pain intensity. It has moderate to good reliability.
RANGE OF MOTION | Baseline and up to one year
  When referring to range of motion, it is understood as the number of degrees through which a joint is capable of moving. To measure the hip, the "Straight Leg Raise Test" (which indirectly measures hamstring extensibility) will be used; hip flexion with the knee flexed (for the gluteus maximus); hip extension using the "Modified Thomas Test" (for the iliopsoas); and hip abduction with the knee extended (for the abductors). At the knee, flexion will be tested with the "Modified Thomas Test," while at the ankle, dorsiflexion will be measured, first with the knee extended using the "Modified Stride Test," and second with the knee flexed using the "Stride Test."
MUSCULAR STRENGTH | Baseline and up to one year
  Isometric muscle strength will be assessed using a dynamometer.